CLINICAL TRIAL: NCT06440187
Title: Phase II Study of Nivolumab Plus Gemcitabine in Patients With Recurrent or Metastatic Nasopharyngeal Carcinoma-HN17-11
Brief Title: Nivolumab Plus Gemcitabine in Patients With Recurrent or Metastatic Nasopharyngeal Carcinoma-HN17-11
Acronym: HN17-11
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Bhumsuk Keam, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KCSG-HN-17-11
Record Dates: First submitted 2018-06-06; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Recurrent or Metastatic Nasopharyngeal Carcinom
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Intervention Model Description: gemcitabine + nivolumab
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- gemcitabine+ nivolumab (Experimental): Nivolumab administration on D1 and D15 every cycle, with 3mg/kg with gmecitabine co-administration on D1 and D15 every cycle, with 1250mg/m2
  Interventions: Drug: Gemcitabine+ nivolumab

INTERVENTIONS:
Drug: Gemcitabine+ nivolumab — Gemcitabine+ nivolumab q 2wks
  Other Names: Experimental group

SUMMARY:
NPC is a highly chemo-sensitive cancer. Platinum-containing doublet chemotherapy is regarded as the standard treatment for patients with recurrent or metastatic NPC, even though it has never been directly compared with supportive care. Until now, no randomized trials have defined the optimum regimens. At present, cisplatin plus continuous intravenous infusion of fluorouracil is widely used in patients with recurrent or metastatic nasopharyngeal carcinoma, with a response rate of 40-65%.

Gemcitabine single is active and tolerable agent for recurred or metastatic NPC. Response rate (RR) was 34% and progression-free survival (PFS) was 5.0 months . Moreover, gemcitabine reduces the frequency of CD11b+GR1+ myeloid suppressor cells. Gemcitabine-induced apoptosis of established tumours may enhance the dendritic cell dependent cross-presentation of tumor antigens to T cells. Gemcitabine can function in synergy with CD40 stimulation of T cells. Hence, theoretically gemcitabine can have synergistic effect with PD-1/PD-L1 blocking agent.

Immunotherapy with immune checkpoint inhibitors has gradually emerged as a promising treatment modality for head and necks squamous cell carcinoma and NPC.

DETAILED DESCRIPTION:
Based on these evidences which suggest a function for PD-1/PD-L1 in NPC and potential synergistic effect with gemcitabine, the use of nivolumab in recurred/metastatic NPC is reasonable and valuable. So we design this phase II study of nivolumab and gemcitabine in recurred/metastatic NPC which is common cancer in Asian.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed nasopharyngeal carcinoma
2. Recurred after local treatment or metastatic disease. Disease that is not amenable to surgery, radiation or combined modality therapy with curative intent
3. Received at least one line of palliative chemotherapy
4. Presence of at least one measurable target lesion for further evaluation according to RECIST 1.1 criteria. Progressive lesions after radiation therapy can also be a target lesion. However, patients who were refractory to initial CCRT with platinum therapy (recurred within 6 months) were excluded.
5. 20 years or older
6. ECOG performance status 0, 1
7. Adequate organ function ANC ≥ 1500/ μL Platelets ≥100,000/ μL Hemoglobin ≥ 9.0 g/dL Serum creatinine ≤1.5 x ULN Serum bilirubin ≤1.5 x ULN AST, ALT, ≤3.0 x ULN (regardless of liver metastasis)
8. A patient with the willingness to comply with the study protocol during the study period and capable of complying with it
9. A patient who signed the informed consent prior to the participation of the study and who understands that he/she has a right to withdrawal from participation in the study at any time without any disadvantages.

Exclusion Criteria:

1. A patient with no measurable disease
2. A patient with previous active or passive immunotherapy or immune check point blocking agents or gemcitabine.
3. Active HBV (HBV DNA is positive) or HCV (HCV RNA is detected) or HIV infection. (inactive HBsAg carrier with prophylactic antiviral treatment can be enrolled)
4. A pregnant or lactating patient
5. A patient of childbearing potential without being tested for pregnancy at baseline or with being tested for positive. (A postmenopausal woman with the amenorrhea period of at least 12 months or longer is considered to have non-childbearing potential)
6. A man or woman of childbearing potential who has no willingness to use a contraceptive measure during the study
7. A patient with history of another malignant disease within past 5 years, except curatively treated basal cell carcinoma of skin, early gastric cancer, and cervical carcinoma in situ.
8. A patient with history of uncontrolled seizures, central nervous system disorder or psychiatric disorders that are considered clinically significant by the investigator that would prohibit the understanding of informed consent or that may be considered to interfere with the compliance of the administration of the study medications.
9. A patient with clinically significant heart disease (e.g. congestive heart failure, symptomatic coronary artery diseases, cardiac arrhythmia, etc) or myocardial infarction within past 12 months.
10. Ongoing cardiac arrhythmia of grade ≥2, atrial fibrillation of any grade, or QTc interval>450msec for males or >470msec for female.
11. A patient with interstitial pneumonia or diffuse symptomatic fibrosis of the lungs
12. A patient with organ transplantation requiring immunosuppressive therapy

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-06-08 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Progression free survival | From the first date of treatment to the date occurring disease progression or death from any cause
  the percentage of patients who have not experienced disease progression or death from any cause from the start of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Seoul National University Hospital, Seoul, South Korea